CLINICAL TRIAL: NCT02353624
Title: Physiological Responses to a Prolonged Cycling Expedition in Older Men
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Professor, University of Copenhagen
Other Study IDs: Nordkapp cycling study
Record Dates: First submitted 2015-01-22; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Aging

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples, muscle and subcutaneous adipose tissue biopsies and venous blood samples.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Cycling — Cycling distance of 2880 km in 14 days

SUMMARY:
The aim of this study was to test the physiological response to a 2800 km cycling expedition, from Copenhagen, Denmark to Nordkapp, Norway, in a group of older male recreational cyclists.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the cycling expedition

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Older male cyclits particpating in the cycling event
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Total daily energy expenditure (Measured using the doubly labeled water technique) | Change from baseline
  Measured using the doubly labeled water technique

SECONDARY OUTCOMES:
Peak fat oxidation (Measured during incremental submaximal exercise) | Change from baseline
  Measured during incremental submaximal exercise

OTHER OUTCOMES:
Energy intake (Measured using selfreported and supervised food logs) | Change from baseline
  Measured using selfreported and supervised food logs
Body composition | Change from baseline
  Measured from isotope dilution
Energy Balance (Discrepancy between energy expenditure and intake or changes in body composition) | Change from baseline
  Discrepancy between energy expenditure and intake or changes in body composition
Cardiac Stress | Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Helge, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen N, Denmark

REFERENCES:
- [Derived] Rosenkilde M, Morville T, Andersen PR, Kjaer K, Rasmusen H, Holst JJ, Dela F, Westerterp K, Sjodin A, Helge JW. Inability to match energy intake with energy expenditure at sustained near-maximal rates of energy expenditure in older men during a 14-d cycling expedition. Am J Clin Nutr. 2015 Dec;102(6):1398-405. doi: 10.3945/ajcn.115.109918. Epub 2015 Oct 21. PMID 26490491